CLINICAL TRIAL: NCT04923204
Title: Genetic Variations Associated With the Therapeutic Response and Profile of Adverse Effects in the Treatment of Bipolar Depression
Brief Title: Utility of the Pharmacogenetic Information Provided by NEUROPHARMAGEN in the Treatment of Bipolar Depressionwith Bipolar Depression
Status: Completed | Type: Observational
Sponsor: AB Biotics, SA (Industry)
Collaborators: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Other Study IDs: PGx-BP
Record Dates: First submitted 2021-05-03; First posted 2021-06-11 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Bipolar Disorder
Keywords: Mood disorders; Pharmacogenomic Testing; Precision Medicine; Adverse events; Treatment response
MeSH Terms: conditions — Bipolar Disorder; Mood Disorders | interventions — Pharmacogenomic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Bipolar depression pharmacogenetics: Patients 18 years and older, with a diagnosis of bipolar disorder with an index episode of depression with or without associated psychotic symptoms (according to the Diagnostic Manual of Mental Disorder 4th Edition Text Revision, DSM-IV-TR), who attended the Bipolar Disorder Program of the Psychiatry Service of the Hospital Clínic de Barcelona (Spain).
  Interventions: Diagnostic Test: Pharmacogenomic-testing with NEUROPHARMAGEN

INTERVENTIONS:
Diagnostic Test: Pharmacogenomic-testing with NEUROPHARMAGEN — This observational retrospective study aims at evaluating the impact of the genetic variation in individual genes on the therapeutic response and side effects profile in a bipolar disorder cohort, using NEUROPHARMAGEN.
  NEUROPHARMAGEN is a pharmacogenomic-based decision support tool that helps clinicians in the selection and dosing of psychoactive drugs based on the integration of pharmacogenetic information.

SUMMARY:
Evaluation of the impact of the genetic variation of individual genes on the therapeutic response and side effects profile in a cohort of well-characterized patients with bipolar depression, using NEUROPHARMAGEN.

DETAILED DESCRIPTION:
Bipolar disorder (BD) is a severe psychiatric condition characterized by mood swings between (hypo)mania and depression, with a total lifetime prevalence of 2.4%. An early and effective therapeutic approach is key for the patient prognosis, being the pharmacotherapy the main therapeutic tool for its management.

Treatment guidelines for BD include a variety of psychotropic medications, including lithium, anticonvulsants, antipsychotics, antidepressants, anxiolytics, and combinations of these medications. However, treatment response is often inadequate and poor tolerability is frequently observed.

Variability in treatment efficacy and tolerability has been shown to be influenced by several factors, including the inherited genetic variation. Several meta-analyses have shown that some genetic variants influence the probability of response to selective serotonin reuptake inhibitors (SSRIs) in patients with depression. Similarly, specific genetic polymorphisms have been associated with the risk of certain antipsychotic-induced adverse effects in patients with schizophrenia. However, the impact of many these variants has not been studied in the context of bipolar disorder.

NEUROPHARMAGEN is a pharmacogenomic-based decision support tool that helps clinicians in the selection and dosing of psychoactive drugs based on the integration of pharmacogenetic information, among other patient's characteristics that influence the medication success.

The clinical utility of NEUROPHARMAGEN has been evaluated in major depression disorder (MDD) through randomized clinical trials with hundreds of patients. Two small pilot trials in bipolar patients have suggested a potential clinical utility of this tool in this patient population. However, the output of pharmacogenomic-based tools such as NEUROPHARMAGEN is based in the analysis of several genes, which could differ in their individual clinical utility in a disorder-related manner.

This observational, retrospective, epidemiological study includes 76 patients who attended the Bipolar Disorder Program of the Psychiatry Service of the Hospital Clinic de Barcelona (Spain) with the aim of objectively evaluate the impact of the genetic variation in individual genes on the therapeutic response and side effects profile in this cohort, using NEUROPHARMAGEN.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Diagnosis of bipolar disorder with an index episode (IE) of depression with or without associated psychotic symptoms, according to the Diagnostic Manual of Mental Disorder 4th Edition Text Revision (DSM-IV-TR)
* Written informed consent to participate in the study
* Attending the Bipolar Disorder Program of the Psychiatry Service of the Hospital Clinic de Barcelona (Spain) for at least 6 months since the beginning of the index episode of the bipolar depression.

Exclusion Criteria:

* Any serious or terminal medical organic disease
* Mental retardation (defined as an intelligence quotient <85)
* Electroconvulsive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who attended the Bipolar Disorder Program of the Psychiatry Service of the Hospital Clinic de Barcelona (Barcelona, Spain) for at least 6 months since the beginning of the index episode of the bipolar depression.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2019-12-05 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression for Bipolar Disorder (CGI-BP-M) | At the time of enrollment (current status after end of index episode)
  The CGI-BP-M is a modified version of the Clinical Global Impression for Bipolar Disorder for the assessment of manic, hypomanic, depressive or mixed symptoms, long-term outcome of bipolar disorder, and the assessment of the efficacy of several treatments. It consists of three subdomains (depression, mania, and overall), each of them with scoring from 1 (normal) to 7 (extremely ill patients).

SECONDARY OUTCOMES:
Hamilton Rating Scale for Depression Rating Scale (HAM-D) | At the time of enrollment (current status after end of index episode)
  HAM-D rates the clinical severity of depression. It has 17 questions, each with three to five possible answers, with scores ranging from 0 to 2 or from 0 to 4, respectively. The total score ranges from 0 to 52 and cut-off scores can be used to classify the depressive disorder.
Functioning Assessment Short Test (FAST) | At the time of enrollment (current status after end of index episode)
  FAST is a brief instrument designed to assess the main functioning problems experienced by psychiatric patients, particularly bipolar patients. It comprises 24 items that assess impairment or disability in six specific areas of functioning: autonomy, occupational functioning, cognitive functioning, financial issues, interpersonal relationships and leisure time. All of items are rated using a 4-point scale (0 = no difficulty, 1 = mild difficulty, 2 = moderate difficulty and 3 = severe difficulty). The global score is obtained by adding up the scores of each item. The higher the score, the more serious the difficulties are.
Clinical Global Impression for Bipolar Disorder (CGI-BP-M) | At onset of index episode (baseline)
  The CGI-BP-M is a modified version of the Clinical Global Impression for Bipolar Disorder for the assessment of manic, hypomanic, depressive or mixed symptoms, long-term outcome of bipolar disorder, and the assessment of the efficacy of several treatments. It consists of three subdomains (depression, mania, and overall), each of them with scoring from 1 (normal) to 7 (extremely ill patients).
Presence of mood switch | Baseline (onset of index episode) to 6 months (or end of the episode)
  Sudden transition from a depressive mood episode to an episode of mania or hypomania.
Number and type of adverse effects | Baseline (onset of index episode) to 6 months (or end of the episode)
  Sociodemographic and clinical data, including the pharmacological treatment in the index episode (IE) and mood switch (the latter for those patients applicable), and the presence and type of side effect associated with the pharmacological treatment in the IE were extracted from all enrolled subjects. The adverse events recorded were as follows: weight gain, dyslipidemia (cholesterol, LDL, HDL, triglycerides), glucose, sedation, extrapyramidal symptoms, seizures, neuroleptic malignant syndrome, corrected QT interval prolongation, sexual dysfunction, and hyperprolactinemia.

CONTACTS AND LOCATIONS:
Overall Officials: Eduard Vieta, MD, PhD, Study Director — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Callegari C, Isella C, Caselli I, Poloni N, Ielmini M. Pharmacogenetic Tests in Reducing Accesses to Emergency Services and Days of Hospitalization in Bipolar Disorder: A 2-Year Mirror Analysis. J Pers Med. 2019 Apr 30;9(2):22. doi: 10.3390/jpm9020022. PMID 31052247
- [Background] Grande I, Berk M, Birmaher B, Vieta E. Bipolar disorder. Lancet. 2016 Apr 9;387(10027):1561-1572. doi: 10.1016/S0140-6736(15)00241-X. Epub 2015 Sep 18. PMID 26388529
- [Background] Han C, Wang SM, Bahk WM, Lee SJ, Patkar AA, Masand PS, Mandelli L, Pae CU, Serretti A. A Pharmacogenomic-based Antidepressant Treatment for Patients with Major Depressive Disorder: Results from an 8-week, Randomized, Single-blinded Clinical Trial. Clin Psychopharmacol Neurosci. 2018 Nov 30;16(4):469-480. doi: 10.9758/cpn.2018.16.4.469. PMID 30466219
- [Background] Ielmini M, Poloni N, Caselli I, Espadaler J, Tuson M, Grecchi A, Callegari C. The utility of pharmacogenetic testing to support the treatment of bipolar disorder. Pharmgenomics Pers Med. 2018 Mar 16;11:35-42. doi: 10.2147/PGPM.S160967. eCollection 2018. PMID 29588611
- [Background] Kato M, Serretti A. Review and meta-analysis of antidepressant pharmacogenetic findings in major depressive disorder. Mol Psychiatry. 2010 May;15(5):473-500. doi: 10.1038/mp.2008.116. Epub 2008 Nov 4. PMID 18982004
- [Background] Kawaguchi DM, Glatt SJ. GRIK4 polymorphism and its association with antidepressant response in depressed patients: a meta-analysis. Pharmacogenomics. 2014 Aug;15(11):1451-9. doi: 10.2217/pgs.14.96. PMID 25303296
- [Background] Lett TA, Wallace TJ, Chowdhury NI, Tiwari AK, Kennedy JL, Muller DJ. Pharmacogenetics of antipsychotic-induced weight gain: review and clinical implications. Mol Psychiatry. 2012 Mar;17(3):242-66. doi: 10.1038/mp.2011.109. Epub 2011 Sep 6. PMID 21894153
- [Background] Mas S, Gasso P, Ritter MA, Malagelada C, Bernardo M, Lafuente A. Pharmacogenetic predictor of extrapyramidal symptoms induced by antipsychotics: multilocus interaction in the mTOR pathway. Eur Neuropsychopharmacol. 2015 Jan;25(1):51-9. doi: 10.1016/j.euroneuro.2014.11.011. Epub 2014 Nov 29. PMID 25499605
- [Background] Menchon JM, Espadaler J, Tuson M, Saiz-Ruiz J, Bobes J, Vieta E, Alvarez E, Perez V. Patient characteristics driving clinical utility in psychiatric pharmacogenetics: a reanalysis from the AB-GEN multicentric trial. J Neural Transm (Vienna). 2019 Jan;126(1):95-99. doi: 10.1007/s00702-018-1879-z. Epub 2018 May 4. PMID 29728861
- [Background] Niitsu T, Fabbri C, Bentini F, Serretti A. Pharmacogenetics in major depression: a comprehensive meta-analysis. Prog Neuropsychopharmacol Biol Psychiatry. 2013 Aug 1;45:183-94. doi: 10.1016/j.pnpbp.2013.05.011. Epub 2013 Jun 1. PMID 23733030
- [Background] Perez V, Salavert A, Espadaler J, Tuson M, Saiz-Ruiz J, Saez-Navarro C, Bobes J, Baca-Garcia E, Vieta E, Olivares JM, Rodriguez-Jimenez R, Villagran JM, Gascon J, Canete-Crespillo J, Sole M, Saiz PA, Ibanez A, de Diego-Adelino J; AB-GEN Collaborative Group; Menchon JM. Efficacy of prospective pharmacogenetic testing in the treatment of major depressive disorder: results of a randomized, double-blind clinical trial. BMC Psychiatry. 2017 Jul 14;17(1):250. doi: 10.1186/s12888-017-1412-1. PMID 28705252
- [Background] Porcelli S, Fabbri C, Serretti A. Meta-analysis of serotonin transporter gene promoter polymorphism (5-HTTLPR) association with antidepressant efficacy. Eur Neuropsychopharmacol. 2012 Apr;22(4):239-58. doi: 10.1016/j.euroneuro.2011.10.003. Epub 2011 Dec 3. PMID 22137564
- [Background] Vilches S, Tuson M, Vieta E, Alvarez E, Espadaler J. Effectiveness of a Pharmacogenetic Tool at Improving Treatment Efficacy in Major Depressive Disorder: A Meta-Analysis of Three Clinical Studies. Pharmaceutics. 2019 Sep 2;11(9):453. doi: 10.3390/pharmaceutics11090453. PMID 31480800